CLINICAL TRIAL: NCT01907737
Title: Combined Brain and Peripheral Nerve Stimulation to Enhance Beneficial Effects of Functional Electrical Stimulation on Hand Motor Function After Stroke
Brief Title: Combined Brain and Peripheral Nerve Stimulation for Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação Faculdade de Medicina (Other)
Responsible Party: Principal Investigator, Adriana Bastos Conforto, Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: P0546/11
Record Dates: First submitted 2013-07-14; First posted 2013-07-25 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active tDCS and active PNS (Active Comparator): 1 session of active transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and active peripheral nerve stimulation (PNS)
  Interventions: Other: Active tDCS; Other: Active PNS
- Active tDCS and sham PNS (Other): 1 session of active transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and sham peripheral nerve stimulation (PNS)
  Interventions: Other: Active tDCS; Other: Sham PNS
- Sham tDCS and active PNS (Other): 1 session of sham transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and active peripheral nerve stimulation (PNS)
  Interventions: Other: Active PNS; Other: Sham tDCS
- Sham tDCS and sham PNS (Sham Comparator): 1 session of sham transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and sham peripheral nerve stimulation (PNS)
  Interventions: Other: Sham tDCS; Other: Sham PNS

INTERVENTIONS:
Other: Active tDCS — Active tDCS will be applied with the anode positioned over the ipsilesional M1 and the cathode over the contralateral supraorbital region for 20 minutes (1mA).
  Arms: Active tDCS and active PNS; Active tDCS and sham PNS
Other: Active PNS — Active PNS will be administered by 2 pairs of surface electrodes (cathode proximal). One pair will overly the median and ulnar nerves at the wrist, and the other pair will overly the radial nerve. Trains of electric stimulation will be delivered at 1 Hz by using isolation units connected to a square pulse stimulator.
  Arms: Active tDCS and active PNS; Sham tDCS and active PNS
Other: Sham tDCS — In sham tDCS, no current will be delivered through the tDCS device.
  Arms: Sham tDCS and active PNS; Sham tDCS and sham PNS
Other: Sham PNS — No current will be delivered to the radial, ulnar and median nerves.
  Arms: Active tDCS and sham PNS; Sham tDCS and sham PNS

SUMMARY:
Cerebrovascular disease is a major cause of disability worldwide. The catastrophic burden of stroke is more dramatic in low- and middle- income countries, and the scarcity of evidence-based rehabilitation interventions represents a major challenge to global health care. Upper limb weakness is frequent after stroke, but there is no universally accepted treatment to effectively improve hand function in patients with moderate and severe motor impairment. These are the patients in deepest need of rehabilitative interventions. This project addresses this important issue, by testing effects of a novel approach. We will non-invasively stimulate the brain and peripheral nerves in order to enhance effects of motor training aided by an electrical stimulation device in patients with moderate to severe hand weakness. Our hypothesis is that brain stimulation, when added to peripheral nerve stimulation, will enhance effects of motor training to a greater extent than brain stimulation alone, peripheral stimulation alone, or no stimulation.

DETAILED DESCRIPTION:
The goal of this study is to compare the effects of FES in close association with either transcranial direct current stimulation (tDCS) alone, peripheral nerve stimulation (PNS)alone, tDCS + PNS or sham tDCS + sham PNS, in patients with moderate to severe upper limb weakness, in a cross-over design. The working hypothesis of this proof-of-principle study is that either tDCS or PNS will enhance effects of functional electrical stimulation (FES) to a greater extent than placebo tDCS and PNS, and that the combination of tDCS and PNS will further improve motor outcomes than either tDCS or PNS alone.

The interventions will consist of outpatient motor training of the paretic wrist with FES in four experimental sessions separated by two weeks. In each session, either active tDCS + sham PNS, active PNS + sham tDCS,active tDCS + active PNS or sham tDCS + sham PNS will be applied. PNS will be applied for 2 hours and tDCS will be applied in the last 20 minutes before completion of PNS. The order of the sessions will be randomized across patients. Before the first session, patients will be familiarized with the FES device.

ELIGIBILITY:
Inclusion Criteria:

* Age, 18 years or older;
* First-ever, ischemic or hemorrhagic stroke at least six months before, confirmed by computed tomography or magnetic resonance imaging;
* Moderate to severe motor impairment of an upper limb, defined as a score between 7 and 50 on the Fugl-Meyer Assessment of Sensorimotor Recovery after stroke, a scale with scores for upper limb ranging from 0 (no function) to 66 (normal function;
* Ability to provide written Informed Consent (patient or legal representative);
* Ability to comply with the schedule of interventions and evaluations in the protocol.

Exclusion Criteria:

* Lack of ability to voluntarily activate any active range of wrist extension;
* Anesthesia of the paretic hand;
* Stroke lesions affecting entirely the hand knob area of the motor cortex120;
* Stroke lesions affecting the cerebellum or the brain stem;
* Severe spasticity at the paretic elbow, wrist, or fingers, defined as a score of >3 on the Modified Ashworth Spasticity Scale;
* Active joint deformity;
* Uncontrolled medical problems such as end-stage cancer or renal disease;
* Pregnancy;
* Seizures;
* Pacemakers;
* Other neurological disorders such as Parkinson's disease;
* Psychiatric illness including severe depression;
* Aphasia or serious cognitive deficits that preclude comprehension of the experimental protocol or ability to provide consent. A score in the Minimental State Examination lower than 23/30 points will be used for patients with higher than 1 year of education, and a score lower than 19/30 will be used for patients with 1 year of education or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Conforto, MD PhD, Principal Investigator — Instituto do Coracao
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo/Fundação Faculdade de Medicina, São Paulo, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- Four Interventions in a Cross-over Design: Each subject participated in four sessions of interventions in different days.
  * 1 session of active transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and active peripheral nerve stimulation (PNS)
  * 1 session of active transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and sham peripheral nerve stimulation (PNS)
  * 1 session of sham transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and active peripheral nerve stimulation (PNS)
  * 1 session of sham transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and sham peripheral nerve stimulation (PNS)
Period: Overall Study
Arm/Group | Four Interventions in a Cross-over Design
Started | 22
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: It was a cross-sectional study. Of twenty two participants who started the study, one participant only participated in one of the four sessions, while the remainder participated in all four. Of the 21 participants who completed four sessions, one was removed from analyses after meeting exclusion criteria
Groups:
- Four Interventions in a Cross-over Design: * 1 session of active transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and active peripheral nerve stimulation (PNS)
  * 1 session of active transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and sham peripheral nerve stimulation (PNS)
  * 1 session of sham transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and active peripheral nerve stimulation (PNS)
  * 1 session of sham transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and sham peripheral nerve stimulation (PNS)
Arm/Group | Four Interventions in a Cross-over Design
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 20

OUTCOME MEASURES:

1. Primary Outcome: Active Range of Motion of Wrist Extension in the Paretic Side
Description: In this cross-over study, the primary outcome was measured immediately before and after each session of treatment. In each session, one of the four possible interventions was administered.
Time Frame: Pre- and post-intervention on each intervention day
Population: Of twenty two participants who started the study, one participant only participated in one of the four sessions, while the remainder participated in all four. Of the 21 participants who completed four sessions, one was removed from analyses after meeting exclusion criteria
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Active tDCS and Active PNS: -1 session of active transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and active peripheral nerve stimulation (PNS)
  Active tDCS and active PNS: Active tDCS will be applied with the anode positioned over the ipsilesional M1 and the cathode over the contralateral supraorbital region for 20 minutes (1mA).
  Active PNS will be administered by 2 pairs of surface electrodes (cathode proximal). One pair will overly the median and ulnar nerves at the wrist, and the other pair will overly the radial nerve. Trains of electric stimulation will be delivered at 1 Hz by using isolation units connected to a square pulse stimulator.
- Active tDCS and Sham PNS: -1 session of active transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and sham peripheral nerve stimulation (PNS)
  Active tDCS and sham PNS: Active tDCS will be applied with the anode positioned over the ipsilesional M1 and the cathode over the contralateral supraorbital region for 20 minutes (1mA). In sham PNS, the median, ulnar and radial nerves will not be actively stimulated.
- Sham tDCS and Active PNS: -1 session of sham transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and active peripheral nerve stimulation (PNS)
  Sham tDCS and active PNS: In sham tDCS, no current will be delivered through the tDCS device. Active PNS will be administered by 2 pairs of surface electrodes (cathode proximal). One pair will overly the median and ulnar nerves at the wrist, and the other pair will overly the radial nerve. Trains of electric stimulation will be delivered at 1 Hz by using isolation units connected to a square pulse stimulator.
- Sham tDCS and Sham PNS: -1 session of sham transcranial direct current stimulation (TDCS) of the hemisphere affected by the stroke and sham peripheral nerve stimulation (PNS)
  Sham tDCS and sham PNS: No current will be delivered by the tDCS device, or to the radial, ulnar and median nerves.
Arm/Group | Active tDCS and Active PNS | Active tDCS and Sham PNS | Sham tDCS and Active PNS | Sham tDCS and Sham PNS
Number analyzed (Participants) | 20 | 20 | 20 | 20
degrees
  Before stimulation | 37.8 (11.6) | 38 (14.2) | 37.2 (13.9) | 38 (14.2)
  After stimulation | 36.5 (13.2) | 36.2 (13.7) | 37.4 (15.1) | 36.2 (13.7)

ADVERSE EVENTS:
Arm/Group | Active tDCS and Active PNS | Active tDCS and Sham PNS | Sham tDCS and Active PNS | Sham tDCS and Sham PNS
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 1/22
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS and Active PNS (N=21) | Active tDCS and Sham PNS (N=21) | Sham tDCS and Active PNS (N=21) | Sham tDCS and Sham PNS (N=22)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The patient reported hip pain while seating during the peripheral stimulation and tDCS sham interventions. 22 subjects were evaluated for adverse events for this session and 21, for the other sessions because this patient only underwent this session

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No